CLINICAL TRIAL: NCT03465670
Title: Clinical Efficacy of Chlorhexidine-based Mouthrinse Formulations in Patients Undergoing Flap Surgery: a Triple Blind, Parallel-arm, Randomized Controlled Trial
Brief Title: Periodontal Wound Healing With CHX and Hyaluronic Acid
Acronym: CHX+HA+ADS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of Ferrara (Other)
Responsible Party: Principal Investigator, Roberto Farina, Full-Time Researcher and Chair of Oral Surgery, University Hospital of Ferrara
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: CHX+HA+ADS
Record Dates: First submitted 2018-03-06; First posted 2018-03-14 (Actual); Last update posted 2018-03-14 (Actual); Status verified 2018-03

CONDITIONS: Surgical Flaps; Wound Healing; Gingiva
Keywords: chlorhexidine; hyaluronic acid; tooth discoloration
MeSH Terms: conditions — Tooth Discoloration

STUDY DESIGN:
Intervention Model Description: Single-center, parallel-arm, triple-blind, randomized controlled clinical trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The patient, the clinical operators as well as the clinical examiner were kept blinded with respect to treatment allocation until the termination of the study. To ensure blindness, CHX and CHX+HA+ADS mouthrinses were provided in identical, masked containers numbered according to the randomization sequence.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CHX (Active Comparator): Post-surgery use of a 0.2% chlorhexidine (CHX) mouthrinse (10 ml for 1 minute, t.i.d. for 21 days)
  Interventions: Device: CHX
- CHX+HA+ADS (Experimental): Post-surgery use of a 0.2% chlorhexidine (CHX) mouthrinse containing 0.2% hyaluronic acid (HA) and Anti-Discoloration System (ADS) (10 ml for 1 minute, t.i.d. for 21 days)
  Interventions: Device: CHX+HA+ADS

INTERVENTIONS:
Device: CHX — Patients received a 21-day supply of 0.2% chlorhexidine (CHX) according to the randomization list, and were instructed to use 10 ml of the assigned mouthrinse for 1 minute, t.i.d. for 21 days. After rinsing, patients were asked to avoid washing their mouth or drinking for 30 minutes. Patients were asked to return the mouthrinse bottles (either empty of filled) at the end of the experimental period (day 21), in order to assess the level of patient compliance with the assigned CHX regimen.
  Arms: CHX
Device: CHX+HA+ADS — Patients received a 21-day supply of 0.2% chlorhexidine (CHX) containing 0.2% hyaluronic acid (HA) and Anti-Discoloration System (ADS) according to the randomization list, and were instructed to use 10 ml of the assigned mouthrinse for 1 minute, t.i.d. for 21 days. After rinsing, patients were asked to avoid washing their mouth or drinking for 30 minutes. Patients were asked to return the mouthrinse bottles (either empty of filled) at the end of the experimental period (day 21), in order to assess the level of patient compliance with the assigned CHX regimen.
  Arms: CHX+HA+ADS

SUMMARY:
Backround: No data on the adjunctive effects of hyaluronic acid (HA) in a post-surgery, chlorhexidine (CHX) - based plaque control regimen are available. Also, contrasting evidence is available regarding the efficacy of CHX-based formulations containing anti-discoloration system (ADS). The aim of the present study was to evaluate the post-surgery gingival healing as well as plaque, gingival inflammation, and staining levels following the use of a 0.2% chlorhexidine (CHX) solution with or without anti-discoloration system (ADS) and 0.2% hyaluronic acid (HA).

Methods: Patients undergoing flap surgery at sites with an intact or reduced but healthy periodontium participated in a parallel-arm RCT. After surgery, patients used the assigned mouthrinse (CHX+HA+ADS or CHX) for 21 days. At day 7 and 21, the Gingival Healing Index (GHI) was used to assess the quality of flap closure at the interdental papilla. Plaque index (PlI), Gingival Index (GI), Angulated bleeding score (AngBS), tooth and tongue staining were also assessed.

ELIGIBILITY:
INCLUSION CRITERIA

Patients were included in the study if positive for each of the following patient related criteria:

* 18 years or older;
* able and willing to provide a written informed consent;
* willing to grant the sufficient compliance with the experimental procedures.

Patients were included in the study if positive for each of the following surgery-related criteria (verified as part of their overall treatment plan):

* indication to at least one session of oral surgery (including periodontal surgery, endodontic surgery, tooth extraction, and implant surgery) requiring the elevation of an envelope or triangular, full-thickness gingival/mucosal flap;
* indication to flap extension to the interdental papilla between either the canine and first premolar or first and second premolar to enhance surgical visibility (teeth in this area were identified as the experimental teeth);
* intact (i.e., no clinical attachment loss) or reduced periodontium with probing pocket depths ≤ 3 mm and no diastema at experimental teeth;
* indication to the repositioning of the surgical flap at the pre-surgical level on the experimental teeth at suturing (i.e. no coronal advancement or apical displacement of the flap).

EXCLUSION CRITERIA

Patients were excluded from the study (at either recruitment or during the experimental phase) if positive for one or more of the following patient-related criteria:

* pregnancy or lactation;
* genetic defects (e.g. Down's syndrome) with an established impact on periodontal status;
* diabetes mellitus;
* immune system disorders (e.g. HIV/AIDS);
* heavy smokers (≥ 10 cigarettes/day);
* severe blood disorders, with a documented qualitative and/or quantitative deficit of polymorphonuclears and/or platelets;
* assumption of medications affecting the gingiva and/or the oral mucosa (e.g. diphenylhydantoin, calcium channel blockers, cyclosporin A, immunostimulants/immunomodulators),
* assumption of oral contraceptives;
* use of systemic or local antibiotics in the previous 4 weeks before study initiation and throughout the entire experimental phase;
* documented allergy to CHX and/or HA.

Patients were excluded from the study if the experimental teeth were positive for one or more of the following criteria:

* dental treatment within the last two months;
* presence of untreated caries or endodontic lesions;
* presence of root fractures;
* tooth alterations (i.e. amelogenesis imperfecta, tetracycline staining) impairing staining evaluations;
* presence of inadequate restorations;
* orthodontic appliances;
* indication to mucogingival surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2015-12-16 (Actual); Primary Completion 2017-06-14 (Actual); Study Completion 2017-06-14 (Actual)

PRIMARY OUTCOMES:
Gingival Healing Index | GHI was evaluated at 7 days following surgery.
  The healing process was evaluated at experimental teeth using a composite index, namely the Gingival Healing Index (GHI), which was created specifically to assess the post-surgery conditions of the interdental papilla. Briefly, the interdental papillae of experimental teeth were visually inspected, and a score was assigned for the severity of wound dehiscence (1-3) and the profile of the buccal and oral aspects of the papilla (1-3). For each patient, GHI score was obtained as the sum of the scores of each variable. Therefore, GHI ranged from 2 (worst quality of healing) to 6 (optimal quality of healing).

SECONDARY OUTCOMES:
Gingival Index (GI) (Löe & Silness 1963) modified by Trombelli et al. (2004) | GI was evaluated immediately before surgery and at 7 and 21 days following surgery.
Angulated bleeding score (AngBs) (van der Weijden et al. 1994) modified by Trombelli et al. (2004) | AngBS was evaluated immediately before surgery and at 7 and 21 days following surgery.
Plaque index (PlI) (Quigley & Hein 1962) modified by Turesky et al. (1970) | PlI was evaluated immediately before surgery and at 7 and 21 days following surgery.
Intensity stain index of Lobene (1968) modified by Grundemann et al. (2000) | Stain Index was evaluated immediately before surgery and at 7 and 21 days following surgery.
Tongue stain (Claydon et al. 2001) | Tongue stain was evaluated immediately before surgery and at 7 and 21 days following surgery.
Gingival Healing Index | GHI was re-evaluated at 21 days following surgery.
  The healing process was evaluated at experimental teeth using a composite index, namely the Gingival Healing Index (GHI), which was created specifically to assess the post-surgery conditions of the interdental papilla. Briefly, the interdental papillae of experimental teeth were visually inspected, and a score was assigned for the severity of wound dehiscence (1-3) and the profile of the buccal and oral aspects of the papilla (1-3). For each patient, GHI score was obtained as the sum of the scores of each variable. Therefore, GHI ranged from 2 (worst quality of healing) to 6 (optimal quality of healing).

CONTACTS AND LOCATIONS:
Locations (1):
- University-Hospital, Ferrara, Italy

IPD SHARING:
Plan to Share IPD: No